CLINICAL TRIAL: NCT07235852
Title: Pilot Testing Into the Feasibility of the Developed Cognitive Behavioral Therapy Intervention
Acronym: CHERISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Keele University (Other); Hayatabad Medical Complex (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KMU/DIR/CTU/2025/007
Record Dates: First submitted 2025-09-26; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Depression; Anxiety Disorders
Keywords: People living with HIV (PLHIV); Cognitive Behavioral Therapy (CBT); Culturally Adapted CBT (Ca-CBT); Feasibility Trial
MeSH Terms: conditions — HIV Infections; Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to one of two parallel arms (Ca-CBT vs Treatment as Usual). Randomization will use central, computer-generated permuted blocks (blocks of 4), administered by an independent researcher.
Who Masked: Outcomes Assessor
Masking Description: Assessors conducting outcome measurements will be blinded to treatment allocation (single-blind design). Randomization and allocation will be performed centrally by an independent researcher not involved in assessments or intervention delivery. Intervention therapists (HIV health workers) and participants will be aware of allocation due to the behavioral nature of the intervention. To reduce accidental unblinding, assessors will be trained to avoid discussing intervention content with participants and will document any instances where they suspect unblinding. Participant perceptions of allocation will be collected post-study to assess potential unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally Adapted Cognitive Behavioral Therapy (Ca-CBT) (Experimental): Participants randomized to this arm will receive a culturally adapted cognitive behavioral therapy (Ca-CBT) intervention delivered by trained HIV health workers. The therapy will consist of six consecutive sessions, each approximately 45-60 minutes, focusing on reducing depression and anxiety symptoms, improving functionality, adherence to antiretroviral therapy (ART), and problem-solving skills. Intervention materials will include culturally relevant stories, metaphors, and self-help audio/video resources, tailored for low-literacy populations.
  Interventions: Behavioral: Culturally Adapted Cognitive Behavioral Therapy (Ca-CBT)
- Treatment as Usual (TAU) (Active Comparator): Participants randomized to this arm will continue to receive routine HIV care as per the HIV Control Program guidelines. This includes free ART initiation and continuation, regular medical check-ups, medication refills, and adherence counselling provided at the Family Care Centre (FCC), Hayatabad Medical Complex, Peshawar. No additional psychological intervention will be provided in this arm.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Culturally Adapted Cognitive Behavioral Therapy (Ca-CBT) — A six-session culturally adapted cognitive behavioral therapy (Ca-CBT) intervention designed for people living with HIV (PLHIV) with depression or anxiety. Sessions will last 45-60 minutes each, delivered weekly by trained HIV health workers under professional supervision. The intervention incorporates culturally relevant stories, metaphors, and self-help audio/video materials, tailored for low-literacy populations. The therapy focuses on reducing depression and anxiety, improving functioning, enhancing adherence to antiretroviral therapy (ART), and problem-solving skills.
  Other Names: Culturally adapted CBT, CaCBT
  Arms: Culturally Adapted Cognitive Behavioral Therapy (Ca-CBT)
Other: Treatment as Usual (TAU) — Participants will receive routine HIV care as provided at Family Care Centres under the National HIV Control Program. This includes free initiation and continuation of antiretroviral therapy (ART), adherence counselling, regular health check-ups, and medication refills. No additional psychological therapy or behavioral intervention will be provided.
  Other Names: Routine HIV care, Standard care under HIV Control Program
  Arms: Treatment as Usual (TAU)

SUMMARY:
This pilot feasibility randomized controlled trial will test a culturally adapted cognitive behavioral therapy (Ca-CBT) intervention for depression and anxiety among people living with HIV (PLHIV) in Peshawar, Pakistan. Fifty participants will be randomized to either receive six sessions of the adapted CBT delivered by trained HIV health workers or treatment as usual (TAU). The study will assess feasibility, acceptability, recruitment and retention rates, and preliminary clinical outcomes, to inform the development of a larger definitive trial.

DETAILED DESCRIPTION:
This feasibility pilot trial aims to evaluate the acceptability and feasibility of a culturally adapted cognitive behavioral therapy (Ca-CBT) intervention for PLHIV with comorbid depression or anxiety in Pakistan. The study will be conducted at the Family Care Centre (FCC), Hayatabad Medical Complex, Peshawar, which provides HIV diagnosis, registration, treatment, and adherence counselling.

Fifty eligible participants aged 18-65, living with HIV, and meeting the Hospital Anxiety and Depression Scale (HADS) thresholds will be randomized (1:1) to intervention or treatment as usual. The intervention group will receive six consecutive sessions of Ca-CBT, designed to improve depression, anxiety, adherence to ART, and functionality. Sessions will use culturally relevant materials, metaphors, and self-help tools, tailored for low-literacy populations. Delivery will be by HIV health workers trained and supervised under a cascade model.

Primary feasibility outcomes include recruitment, retention, completion of therapy sessions, fidelity of delivery, and acceptability. Secondary outcomes include changes in depression (HADS), functioning (WHODAS), internalized stigma, ART adherence self-efficacy, health-related quality of life (EQ-5D), and trauma symptoms. Assessments will occur at baseline, 8 weeks (post-intervention), and 12 weeks (follow-up).

The trial uses a randomized, single-blind (assessors) two-arm design. Recruitment will draw from the FCC registry of HIV patients. Sample size justification follows CONSORT guidelines for feasibility trials, with traffic-light progression criteria (stop/amend/go thresholds) for decision-making on a definitive trial.

This study will provide essential data on feasibility, acceptability, and preliminary clinical signals to inform a full-scale RCT evaluating culturally adapted CBT for PLHIV in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Pakistani nationals and residents.
* Confirmed HIV diagnosis (newly diagnosed or on ART within 1 month of diagnosis, or already on lifelong ART, according to UNAIDS HIV diagnostic standards).
* Meeting criteria for depression and anxiety: HADS subscale score >8 on both depression and anxiety, and total HADS score >15.
* HIV patients with comorbid conditions (e.g., Hepatitis, HCV) may be included if HIV is the primary condition.

Exclusion Criteria:

* Diagnosis of bipolar disorder, psychosis, or other severe mental illness according to ICD-11 or DSM-5-TR.
* Evidence of learning disability or severe substance use disorder (except nicotine).
* Currently receiving psychotherapy or antidepressant medication within the last 6 months.
* Current suicidality (per WHO mhGAP) or suicide attempt within the last 2 years.
* HIV-associated neurocognitive disorders (HAND) or severe complications of HIV preventing participation, as judged by treating physician.
* Living in the same household as another study participant (to prevent contamination between arms).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Recruitment - Enrollment Rate | Baseline to 12 weeks post-intervention.
  The proportion of eligible participants who are successfully enrolled into the trial. This will be calculated as: (Number of participants enrolled / Number of eligible participants screened) * 100%.
  Criteria: Proportion completing outcome assessments at 12 weeks (stop <60%, amend 60-80%, go >80%).
Feasibility of Intervention - Retention in Therapy | At the end of the 6-week intervention period
  The proportion of enrolled participants who complete at least 4 out of the 6 planned therapy sessions. This will be calculated as: (Number of participants completing ≥4 sessions / Total number of participants enrolled in the intervention arm) * 100%.
  Criteria: proportion completing outcome assessments at 12 weeks (stop <60%, amend 60-80%, go >80%).
  Go: >80%
Feasibility of Data Collection - Follow-up Assessment Completion | 12 weeks post-intervention
  The proportion of enrolled participants who complete the primary outcome assessments at the 12-week post-intervention time point. This will be calculated as: (Number of participants completing the 12-week assessment / Total number of participants enrolled) * 100%.
  Criteria: proportion completing outcome assessments at 12 weeks (stop <60%, amend 60-80%, go >80%).
  Go: >80%

SECONDARY OUTCOMES:
Change in depression and anxiety symptoms | Baseline, 8 weeks, and 12 weeks.
  Measured using the Hospital Anxiety and Depression Scale (HADS). Each subscale (anxiety & depression) ranges 0-21; higher scores = worse symptoms. Cutoff: ≥8 = probable case. Total score 0-42.
Change in functioning | Baseline, 8 weeks, 12 weeks.
  Measured using the WHO Disability Assessment Schedule (WHODAS 2.0, 12-item). Scores are summed and transformed to 0-100, with higher scores = greater disability / worse functioning.
Change in internalized stigma | Baseline, 8 weeks, 12 weeks.
  Measured using the Brief Internalized Stigma of Mental Illness Scale (ISMI-10). Items scored 1-4, total range 10-40; higher scores = greater stigma.
Change in ART adherence self-efficacy | Baseline, 8 weeks, 12 weeks.
  Measured using the HIV Adherence Self-Efficacy Scale (HIV-ASES). Items rated 1-10; higher scores = greater self-efficacy for ART adherence.
Change in health-related quality of life | Baseline, 8 weeks, 12 weeks.
  Measured using the EuroQol EQ-5D (5 domains, scored 1-3 or 1-5 depending on version; converted to index values 0 = death, 1 = perfect health; higher = better HRQoL). Includes EQ-VAS (0-100 scale).
Change in trauma symptoms | Baseline, 8 weeks, 12 weeks.
  Measured using the Harvard Trauma Questionnaire (HTQ). Items scored 1-4; mean score ≥2.5 suggests clinically significant PTSD symptoms. Higher scores = worse trauma symptoms.
Intervention fidelity | Baseline, 8 weeks, 12 weeks.
  Measured using the Revised Cognitive Therapy Scale (CTS-R). Each item scored 0-6; total mean score ≥3 indicates adequate competence.
Acceptability of intervention | Baseline, 8 weeks, 12 weeks.
  Measured using the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM). Each tool has 4 items scored 1-5; higher scores = greater acceptability, appropriateness, or feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Mughal, MPH,PhD*, Principal Investigator — Keele University; Prof Monica Magadi, PhD, Principal Investigator — Keele University; Dr James Prior, PhD, Principal Investigator — Keele University; Prof Saeed Farooq, PhD, Principal Investigator — Keele University; Dr Shaista Rasool, PhD, Principal Investigator — Khyber Medical University; Dr Mirat Gul, PhD, Principal Investigator — Mayo Hospital Lahore
Locations (1):
- Family Care Centre (FCC), Hayatabad Medical Complex, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The Individual Participant Data (IPD) from this pilot feasibility trial will be shared with qualified researchers upon request. The dataset will include anonymized data on participant demographics, eligibility, baseline measures, outcome assessments (HADS, WHODAS, ISMI, HIV-ASES, etc.), and data related to the intervention (Ca-CBT or Treatment as Usual). The data sharing plan ensures that participant confidentiality is maintained in accordance with ethical standards, and the dataset will be accessible for further analyses related to mental health interventions for HIV-positive individuals.
  Data sharing will also be contingent upon institutional approval and the availability of resources for analysis. Access will be governed by ethical review board policies to protect participant privacy and confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: he anonymized IPD will be made available within 6 months after the final study results have been published or upon completion of the trial's final analysis. The data will be shared for a minimum of 5 years after study completion for continued scientific exploration.
Access Criteria: Researchers wishing to access the data will need to submit a request to the Principal Investigator or Study Coordinator. Data will be provided to individuals and institutions with ethical approval from an Institutional Review Board (IRB) or Ethics Committee (EC), ensuring adherence to all confidentiality and privacy guidelines. Access will be provided under terms of a data use agreement (DUA) to guarantee appropriate and responsible use of the data.

REFERENCES:
- [Background] Anand S, Hanson K. Disability-adjusted life years: a critical review. J Health Econ. 1997 Dec;16(6):685-702. doi: 10.1016/s0167-6296(97)00005-2. PMID 10176779
- [Background] Benish SG, Quintana S, Wampold BE. Culturally adapted psychotherapy and the legitimacy of myth: a direct-comparison meta-analysis. J Couns Psychol. 2011 Jul;58(3):279-89. doi: 10.1037/a0023626. PMID 21604860
- [Background] Ciesla JA, Roberts JE. Meta-analysis of the relationship between HIV infection and risk for depressive disorders. Am J Psychiatry. 2001 May;158(5):725-30. doi: 10.1176/appi.ajp.158.5.725. PMID 11329393
- [Background] Chowdhary N, Jotheeswaran AT, Nadkarni A, Hollon SD, King M, Jordans MJ, Rahman A, Verdeli H, Araya R, Patel V. The methods and outcomes of cultural adaptations of psychological treatments for depressive disorders: a systematic review. Psychol Med. 2014 Apr;44(6):1131-46. doi: 10.1017/S0033291713001785. Epub 2013 Jul 19. PMID 23866176
- [Background] Degnan A, Baker S, Edge D, Nottidge W, Noke M, Press CJ, Husain N, Rathod S, Drake RJ. The nature and efficacy of culturally-adapted psychosocial interventions for schizophrenia: a systematic review and meta-analysis. Psychol Med. 2018 Apr;48(5):714-727. doi: 10.1017/S0033291717002264. Epub 2017 Aug 23. PMID 28830574
- [Background] Eldridge SM, Ashby D, Kerry S. Sample size for cluster randomized trials: effect of coefficient of variation of cluster size and analysis method. Int J Epidemiol. 2006 Oct;35(5):1292-300. doi: 10.1093/ije/dyl129. Epub 2006 Aug 30. PMID 16943232
- [Background] Hodge DR, Jackson KF, Vaughn MG. Culturally sensitive interventions and health and behavioral health youth outcomes: a meta-analytic review. Soc Work Health Care. 2010;49(5):401-23. doi: 10.1080/00981381003648398. PMID 20521205
- [Background] Huey SJ Jr, Polo AJ. Evidence-based psychosocial treatments for ethnic minority youth. J Clin Child Adolesc Psychol. 2008 Jan;37(1):262-301. doi: 10.1080/15374410701820174. PMID 18444061
- [Background] Li W, Zhang L, Luo X, Liu B, Liu Z, Lin F, Liu Z, Xie Y, Hudson M, Rathod S, Kingdon D, Husain N, Liu X, Ayub M, Naeem F. A qualitative study to explore views of patients', carers' and mental health professionals' to inform cultural adaptation of CBT for psychosis (CBTp) in China. BMC Psychiatry. 2017 Apr 8;17(1):131. doi: 10.1186/s12888-017-1290-6. PMID 28390407
- [Background] Lloyd KR, Jacob KS, Patel V, St Louis L, Bhugra D, Mann AH. The development of the Short Explanatory Model Interview (SEMI) and its use among primary-care attenders with common mental disorders. Psychol Med. 1998 Sep;28(5):1231-7. doi: 10.1017/s0033291798007065. PMID 9794030
- [Background] Mir F, Mahmood F, Siddiqui AR, Baqi S, Abidi SH, Kazi AM, Nathwani AA, Ladhani A, Qamar FN, Soofi SB, Memon SA, Soomro J, Shaikh SA, Simms V, Khan P, Ferrand RA. HIV infection predominantly affecting children in Sindh, Pakistan, 2019: a cross-sectional study of an outbreak. Lancet Infect Dis. 2020 Mar;20(3):362-370. doi: 10.1016/S1473-3099(19)30743-1. Epub 2019 Dec 19. PMID 31866326
- [Background] van Loon A, van Schaik A, Dekker J, Beekman A. Bridging the gap for ethnic minority adult outpatients with depression and anxiety disorders by culturally adapted treatments. J Affect Disord. 2013 May;147(1-3):9-16. doi: 10.1016/j.jad.2012.12.014. Epub 2013 Jan 23. PMID 23351566